CLINICAL TRIAL: NCT01009775
Title: A Phase II, Multicenter, Open-Label Study Of YM155 Plus Docetaxel in Subjects With Stage III (Unresectable) or Stage IV Melanoma
Brief Title: A Study of YM155 Plus Docetaxel in Subjects With Stage III (Unresectable) or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155-CL-034; 2009-015738-31 (EudraCT Number)
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-08

CONDITIONS: Melanoma
Keywords: Melanoma, Stage III; Melanoma, Stage IV; YM 155; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — sepantronium; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM155 plus docetaxel (Experimental)
  Interventions: Drug: YM155; Drug: Docetaxel

INTERVENTIONS:
Drug: YM155 — intravenous infusion
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere

SUMMARY:
The purpose of the study is to evaluate survival, response rate, safety and tolerability of YM155 given in combination with docetaxel in subjects with Stage III (unresectable) and Stage IV melanoma.

DETAILED DESCRIPTION:
All subjects will receive YM155 and docetaxel given in a 21-day cycle. The docetaxel dose will be established based on the findings of the lead-in portion of the study (Part 1). Once the docetaxel dose is established, Part 2 enrollment will begin.

Part 1:

Part 1 is a lead-in stage that will confirm if YM155 can be safely administered in combination with docetaxel at a specified dose.

Part 2:

Subjects enrolled in Part 2 will receive YM155 and docetaxel at the dose established during Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage III (unresectable) or Stage IV melanoma
* No prior systemic treatment or Cytotoxic chemotherapy for advanced melanoma (Stage III or Stage IV)
* If the subject is female, she must be non-pregnant and non-lactating at the Baseline Visit. All sexually active males and females of childbearing potential must agree to use an adequate method of contraception throughout the study period
* Eastern Cooperative Oncology Group (ECOG) performance status </= 1
* Life expectancy > 12 weeks
* At least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors ({RECIST} version 1.1)
* Subjects with a previous history of non-melanoma malignancy must have undergone curative therapy for all prior malignancies and be considered disease free for at least 5 years

Exclusion Criteria:

* Major surgery within 21 days of the Baseline Visit
* Presence or history of brain metastases
* Primary ocular, choroidal or mucosal melanoma
* Known history of positive test for Hepatitis B surface Antigen (HsbAg) or Hepatitis C antibody or history of positive test for Human Immunodeficiency Virus (HIV)
* Hypersensitivity to docetaxel or polysorbate 80
* Neuropathy greater than or equal to Grade 2 at Baseline Visit
* The subject has been previously treated with YM155
* Inadequate marrow, hepatic, and/or renal functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
6-month Progression-free survival | After the last non-progressing subject completes 6 months or discontinues the treatment

SECONDARY OUTCOMES:
Objective response rate (proportion of subjects with complete response or partial response) | After the last non-progressing subject completes 6 months or discontinues the treatment
1 year survival | After the last non-progressing subject completes 6 months or discontinues the treatment
Overall survival | 2 years after the last subject discontinues treatment
Duration of response | After the last non-progressing subject completes 6 months or discontinues the treatment
Clinical benefit rate | After the last non-progressing subject completes 6 months or discontinues the treatment
Time to response | After the last non-progressing subject completes 6 months or discontinues the treatment
Safety assessed by recording of adverse events, physical examinations, vital signs, laboratory assessments and electrocardiograms (ECGs) | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development
Locations (11):
- United States (10):
  - University of South Alabama, Mobile, Alabama
  - Arizona Clinical Research Center, Tuscon, Arizona
  - The Angeles Clinic and Research, Los Angeles, California
  - UCLA, Los Angeles, California
  - Redwood Regional Medical Group, Sebastopol, California
  - University of Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Univ. of Michigan Health System, Ann Arbor, Michigan
  - St. Lukes Hospital Cancer Center, Bethlehem, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- London Regional Cancer Centre, London, Ontario, Canada